CLINICAL TRIAL: NCT05900622
Title: A Study of Modified Limb Braking and Early Bed Mobility Strategies After Femoral Venipuncture Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tong Zhu (Other)
Responsible Party: Sponsor-Investigator, Tong Zhu, Chief physician，Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2023]23th
Record Dates: First submitted 2023-05-23; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Deep Vein Thrombosis; Deep Venous Insufficiency
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Lower extremity on the puncture side with a 4-hour brake+Get out of bed after 8 hours
- Test group A (Experimental): Lower extremity on the puncture side with a 2-hour brake+Get out of bed after 4 hours
  Interventions: Other: Reduced postoperative braking and bed rest time.Lower extremity on the puncture side with a 2-hour brake+Get out of bed after 4 hours
- Test group B (Experimental): No braking of the lower limb on the side of the puncture+Get out of bed after 2 hours
  Interventions: Other: Significantly reduce postoperative braking and bed rest time.No braking of the lower limb on the side of the puncture+Get out of bed after 2 hours

INTERVENTIONS:
Other: Reduced postoperative braking and bed rest time.Lower extremity on the puncture side with a 2-hour brake+Get out of bed after 4 hours — Braking time is defined as the time from the start of postoperative lying down until the patient sits up in bed and can move the lower limbs Bed rest is the time from when the patient is lying down to when they are on the floor after the procedure, but it has been identified as the most difficult part of post-vascular puncture intervention care
  Arms: Test group A
Other: Significantly reduce postoperative braking and bed rest time.No braking of the lower limb on the side of the puncture+Get out of bed after 2 hours — Braking time is defined as the time from the start of postoperative lying down until the patient sits up in bed and can move the lower limbs Bed rest is the time from when the patient is lying down to when they are on the floor after the procedure, but it has been identified as the most difficult part of post-vascular puncture intervention care
  Arms: Test group B

SUMMARY:
The goal of this clinical trial is to compare in describe participant population health conditions. The main questions it aims to answer are:

* To obtain the limb movement and bed mobility limits after femoral venipuncture, in order to provide a basis and support for clinical reduction of postoperative braking time and alleviation of postoperative patient subjective discomfort
* To analyze the effect of perioperative factors such as anticoagulation and sheath size on the complication rate, so as to develop a detailed and systematic strategy to stop bleeding after femoral venipuncture
* The advantages and necessity of reducing the postoperative braking time in bed were demonstrated by objective evaluation of patients' postoperative subjective feelings and mental status.

In this prospective study, 150 patients who underwent femoral vein puncture intervention were selected by inclusion and exclusion criteria, and were randomly divided into control group, trial A group and trial B group by SPSS software, with 50 cases each. In the control group, the lower limb of the punctured side was braked for 4 hours + 8 hours after routine postoperative activities; in the trial A group, the lower limb of the punctured side was braked for 2 hours + 4 hours after postoperative activities; in the trial B group, the lower limb of the punctured side was braked for no postoperative activities + 2 hours after postoperative activities, and the corresponding evaluation indexes and questionnaires were used to record the hemostasis at the puncture site, whether complications occurred and the subjective feelings of patients in each group after completing the corresponding strategies. The data were also recorded along with the general information of the patients and the factors that may cause bleeding in the perioperative period. Statistical analysis was used to classify, summarize and draw conclusions about the data obtained, analyze the limit of braking bed time, and formulate scientific hemostatic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, no serious liver or kidney function abnormalities.
* No significant preoperative bleeding tendency or hemostatic dysfunction, platelets ≥75×109/L, prothrombin time (PT) <16 s.
* No other femoral vascular puncture procedures were performed bilaterally during the observation period.
* Normal neurological and cognitive function, able to make a correct assessment, able to move normally on the floor after surgery, informed consent and willing to cooperate.

Exclusion Criteria:

* Patients in whom this operation is combined with ipsilateral femoral artery puncture or intraoperative percutaneous puncture into the femoral artery by mistake.
* Patients with significant hematoma during femoral vein puncture or with the formation of a visually visible hematoma at the puncture site after removal of the sheath or persistent blood leakage, pseudoaneurysm, or arteriovenous fistula.
* Patients with severe insufficiency of important organs or obvious hemostasis and coagulation dysfunction.
* Patients with poor postoperative compliance or other insurmountable reasons for inability to complete the prescribed time of activity and get out of bed.
* Patients who are unwilling to sign the informed consent form after being adequately informed by the investigator about the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Degree of postoperative bleeding | 8 hours after surgery
  he Christenson modification method [13 was applied to classify the degree of bleeding into normal, non-significant bleeding, and significant bleeding. (1) Normal: no visible bloody exudate on the dressing; (2) Non-significant bleeding: a small amount of localized bleeding, no palpable hematoma or hematoma <5 cm, no special treatment required; (3) Significant bleeding: more bleeding from the dressing, estimated bleeding volume >100 ml, hematoma and skin petechiae >5 cm in diameter, hematoma compression affecting dorsalis pedis artery pulsation, requiring manual compression, sandbag compression or re Compression dressing

SECONDARY OUTCOMES:
Postoperative pain level | 6 hours after surgery
  The numeric rating scale (NRS) was used to assess the pain level of each group of patients from 4 to 6 h after surgery. 0 indicates no pain, 1 to 3 indicates mild pain, 4 to 6 indicates moderate pain, 7 to 9 indicates severe pain, and 10 indicates severe pain, which was rated by patients based on subjective feelings.
Postoperative anxiety level | 6 hours after surgery
  The Hamilton Anxiety Scale (HAMA) was used to assess the anxiety level of each group of patients at 4-6 h postoperatively. A HAMA score of <7 indicates no anxiety, ≥7 indicates possible anxiety, ≥14 indicates definite anxiety, ≥21 indicates definite significant anxiety, and ≥29 indicates severe anxiety.
Postoperative comfort level | 6 hours after surgery
  The kolcaba Comfort Questionnaire (GCQ) was used to assess the comfort level of each group of patients at 4-6 h postoperatively. The higher the GCQ score, the better the comfort level.

IPD SHARING:
Plan to Share IPD: No